CLINICAL TRIAL: NCT06465706
Title: A Prospective, Multicenter, Randomized Controlled Trial Assessing the Safety and Efficacy of the LAmbre™ Plus Left Atrial Appendage Closure System to REDUCE the Risk of Thromboembolism in Patients With Non-Valvular Atrial Fibrillation
Brief Title: Assessing the Safety and Efficacy of the LAmbre™ Plus Device
Acronym: REDUCE-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LA-US-01
Record Dates: First submitted 2024-06-10; First posted 2024-06-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation
Keywords: Left Atrial Appendage Occlusion; Stroke Risk
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients and family will be blinded to which device they received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LAmbre Device (Experimental): LAmbre Plus LAAO is a second-generation device intended for investigational use only in the United States.
  Interventions: Device: LAmbre investigational device
- FDA approved LAAO devices (Active Comparator): The control devices for the study will be commercially available transcatheter LAAO devices. Currently, there are three FDA approved devices (WATCHMAN FLX and WATCHMAN FLX Pro from Boston Scientific and Amplatzer Amulet from Abbott Laboratories) all of which can be used in subjects assigned to the control group.
  Interventions: Device: LAmbre investigational device

INTERVENTIONS:
Device: LAmbre investigational device — Randomized 1:1 to either experimental group or control group.

SUMMARY:
Randomized controlled trial assessing the safety and efficacy of the LAmbre Plus LAA Closure System to rescue the risk of thromboembolism in patients with non-valvular AF.

DETAILED DESCRIPTION:
The goal of this clinical trial is to demonstrate the safety and efficacy of the LAmbre Plus device in patients with non-valvular atrial fibrillation in comparison with the commercially available transcatheter LAAO device(s). The main questions it aims to answer are:

Overall safety of the device that is assessed at the 12 month time period. Overall efficacy, after all subjects have reached the 18 month time period.

Participants will be randomized to either the LAmbre device or other FDA approved LAAO devices.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male or non-pregnant female ≥18 years of age
* The patient has documented paroxysmal, persistent, or permanent non- valvular atrial fibrillation
* The patient has a CHADS2 score ≥ 2 or a CHA2DS2-VASc score of ≥ 3, and is recommended for oral anticoagulation therapy
* The patient is deemed by their physician to be suitable for short-term warfarin therapy, but there is an appropriate rationale for seeking a non-pharmacologic alternative to oral anticoagulation
* The patient is deemed suitable for LAA closure by a multidisciplinary heart team, including at least 1 investigator (e.g. cardiologists) and 1 clinician not involved as part of the procedure team using a shared decision making process, and this determination has been documented in the patient's medical record
* The patient is willing and able to comply with protocol-specified treatment and follow-up evaluations
* The patient (or his or her legally authorized representative) has been informed of the nature of the study, agrees to its provisions, and has been provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

Exclusion Criteria:

* Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure. Female patients of childbearing potential must have a negative pregnancy test done within 7 days prior to index procedure per site standard test.
* Patients with atrial fibrillation that is defined by a single occurrence, or that is transient or reversible (e.g., secondary to CABG, an interventional procedure, pneumonia, or hyperthyroidism)
* Patients who require long-term anticoagulation for a condition other than atrial fibrillation
* Patients with an indication for chronic P2Y12 platelet inhibition therapy
* Patients not suitable for short term warfarin (including due to bleeding diathesis or coagulopathy or absolute contraindication warfarin) or who will refuse transfusion
* Patients with rheumatic mitral valve disease, known severe aortic stenosis requiring surgical or percutaneous valve replacement, or existing mechanical valve prosthesis
* Active infection with bacteremia
* Known hypersensitivity or contraindication to aspirin, clopidogrel, heparin/bivalirudin, any device material or component (nitinol, nickel, titanium, PET), and/or contrast sensitivity that cannot be adequately pre-medicated
* Anatomic conditions that would prevent performance of the LAA occlusion procedure (e.g., prior atrial septal defect [ASD] or patient foramen ovale [PFO] surgical repair or implanted closure device, or obliterated left atrial appendage)
* Recent (within 30 days pre-procedure) or planned (within 60 days post- procedure) cardiac or non-cardiac interventional or surgical procedure (e.g., cardioversion, ablation, percutaneous coronary intervention, cataract surgery, etc.)
* Recent (within 90 days pre-procedure) stroke, transient ischemic attack, or myocardial infarction
* Severe heart failure (New York Heart Association Class IV)
* Known asymptomatic carotid artery disease with>70% diameter stenosis OR symptomatic carotid disease (>50% diameter stenosis with ipsilateral stroke or TIA). Subjects with prior carotid endarterectomy or carotid stent placement may be enrolled, provided that known diameter stenosis is <50%.
* Past or pending heart or any other organ transplant, or on the waiting list for any organ transplant
* Known other medical illness or known history of substance abuse that may cause non-compliance with the protocol, confound data interpretation, or is associated with a life expectancy of less than 2 years
* Current participation in another investigational drug or device study Echocardiographic Exclusion Criteria
* Left atrial appendage anatomy cannot accommodate either the LAmbre Plus LAAO device or the Control device per manufacturer IFU (e.g., the anatomy and sizing must be for both device to be enrolled in the trial or maximum LAAO length < maximum ostium width by TEE)
* LVEF <30%
* Intracardiac thrombus or dense spontaneous echo contrast, as visualized by TEE within 2 days prior to implant
* Moderate or large circumferential pericardial effusion >10 mm or symptomatic pericardial effusion, signs or symptoms of acute or chronic pericarditis, or evidence of tamponade physiology. In the event of a treatable pericardial effusion, the subject may undergo implantation at a later time after it is adequately treated.
* Atrial septal defect that warrants closure.
* Presence of a high risk patent foramen ovale (PFO), defined as an atrial septal aneurysm (excursion >15 mm or length >15 mm) or large shunt (early, within 3 beats and/or substantial passage of bubbles)
* Moderate or severe mitral valve stenosis (mitral valve area <1.5 cm2)
* Complex atheroma with mobile plaque of the descending aorta and/or aortic arch (Grade 4 or higher)
* Evidence of a Cardiac Tumor

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1826 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Major procedure related complications - cardiac perforation | up to 7 days following implant procedure
  Cardiac perforation can be seen interprocedurally through ICE or TEE, post procedurally via TTE or TEE.
Major procedure related complications - pericardial effusion with tamponade or requiring drainage | up to 7 days following implant procedure
  Common complications can be seen interprocedurally through ICE or TEE, post procedurally via TTE or TEE.
Major procedure related complications - device embolization | up to 7 days following implant procedure
  Procedure complications can be seen interprocedurally through ICE or TEE, post procedurally via TTE or TEE.
Major adverse event - Death | up to 7 days following implant procedure
  Death is observed by lack of oxygen, lack of pulse, succession of neurological activity.
Major adverse event - all strokes | up to 7 days following implant procedure
  Stroke is identified by neurologic imaging and transient or permanent motor or sensory deficient.
Major adverse event - systemic embolization | up to 7 days following implant procedure
  Systemic embolization assessed by onsite symptoms and confirmed by diagnostic imaging.
Major adverse event - major bleeding | up to 7 days following implant procedure
  Visual bleeding or a drop in hemoglobin of 2 units and requiring transfusion.

SECONDARY OUTCOMES:
Major adverse event | 45 days, 6 months, 12 months, 18 months and 2, 3, 4, and 5 years
  composite of cardiovascular death, overs CNS injury and major bleeding
mortality | 45 days, 6 months, 12 months, 18 months and 2, 3, 4, and 5 years
  cardiovascular or non-cardiovascular and reported cumulatively and individually
myocardial infarction | 45 days, 6 months, 12 months, 18 months and 2, 3, 4, and 5 years
  Defined as ST or nonST ECG changes with positive cardiac bio markers.
periprocedural stroke | 45 days, 6 months, 12 months, 18 months and 2, 3, 4, and 5 years
  Motor and sensory deficits observed and imaging confirmed.
bleeding complications | 45 days, 6 months, 12 months, 18 months and 2, 3, 4, and 5 years
  Visual bleeding or a drop in hemoglobin
major procedure-related complications | 45 days, 6 months, 12 months, 18 months and 2, 3, 4, and 5 years
  vascular or cardiac complications occurring due to the procedure.
vascular complications | 45 days, 6 months, 12 months, 18 months and 2, 3, 4, and 5 years
  vascular complications are hematomas, aneurysms, and ischemic limb.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — KCCARF

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lansky AJ, Messe SR, Brickman AM, Dwyer M, van der Worp HB, Lazar RM, Pietras CG, Abrams KJ, McFadden E, Petersen NH, Browndyke J, Prendergast B, Ng VG, Cutlip DE, Kapadia S, Krucoff MW, Linke A, Moy CS, Schofer J, van Es GA, Virmani R, Popma J, Parides MK, Kodali S, Bilello M, Zivadinov R, Akar J, Furie KL, Gress D, Voros S, Moses J, Greer D, Forrest JK, Holmes D, Kappetein AP, Mack M, Baumbach A. Proposed Standardized Neurological Endpoints for Cardiovascular Clinical Trials: An Academic Research Consortium Initiative. J Am Coll Cardiol. 2017 Feb 14;69(6):679-691. doi: 10.1016/j.jacc.2016.11.045. PMID 28183511
- [Background] Mandalenakis Z, Von Koch L, Eriksson H, Dellborg M, Caidahl K, Welin L, Rosengren A, Hansson PO. The risk of atrial fibrillation in the general male population: a lifetime follow-up of 50-year-old men. Europace. 2015 Jul;17(7):1018-22. doi: 10.1093/europace/euv036. Epub 2015 Apr 4. PMID 25842274
- [Background] Kalmykov NP, Mashchenko EN. New data on the migration of the family Elephantidae (Mammalia, Proboscidea) in Eurasia. Dokl Biol Sci. 2006 Jan-Feb;406:103-5. doi: 10.1134/s0012496606010303. No abstract available. PMID 16572828
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Dewland TA, Olgin JE, Vittinghoff E, Marcus GM. Incident atrial fibrillation among Asians, Hispanics, blacks, and whites. Circulation. 2013 Dec 3;128(23):2470-7. doi: 10.1161/CIRCULATIONAHA.113.002449. Epub 2013 Oct 8. PMID 24103419
- [Background] Lau DH, Nattel S, Kalman JM, Sanders P. Modifiable Risk Factors and Atrial Fibrillation. Circulation. 2017 Aug 8;136(6):583-596. doi: 10.1161/CIRCULATIONAHA.116.023163. PMID 28784826
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Background] Stewart S, Hart CL, Hole DJ, McMurray JJ. A population-based study of the long-term risks associated with atrial fibrillation: 20-year follow-up of the Renfrew/Paisley study. Am J Med. 2002 Oct 1;113(5):359-64. doi: 10.1016/s0002-9343(02)01236-6. PMID 12401529
- [Background] Al-Saady NM, Obel OA, Camm AJ. Left atrial appendage: structure, function, and role in thromboembolism. Heart. 1999 Nov;82(5):547-54. doi: 10.1136/hrt.82.5.547. PMID 10525506
- [Background] Kong B, Liu Y, Huang H, Jiang H, Huang C. Left atrial appendage closure for thromboembolism prevention in patients with atrial fibrillation: advances and perspectives. J Thorac Dis. 2015 Feb;7(2):199-203. doi: 10.3978/j.issn.2072-1439.2015.01.20. PMID 25713737
- [Background] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Gage BF, van Walraven C, Pearce L, Hart RG, Koudstaal PJ, Boode BS, Petersen P. Selecting patients with atrial fibrillation for anticoagulation: stroke risk stratification in patients taking aspirin. Circulation. 2004 Oct 19;110(16):2287-92. doi: 10.1161/01.CIR.0000145172.55640.93. Epub 2004 Oct 11. PMID 15477396
- [Background] Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest. 2010 Feb;137(2):263-72. doi: 10.1378/chest.09-1584. Epub 2009 Sep 17. PMID 19762550
- [Background] Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010 Nov;138(5):1093-100. doi: 10.1378/chest.10-0134. Epub 2010 Mar 18. PMID 20299623
- [Background] Chan PS, Maddox TM, Tang F, Spinler S, Spertus JA. Practice-level variation in warfarin use among outpatients with atrial fibrillation (from the NCDR PINNACLE program). Am J Cardiol. 2011 Oct 15;108(8):1136-40. doi: 10.1016/j.amjcard.2011.06.017. Epub 2011 Jul 26. PMID 21798501
- [Background] Brass LM, Krumholz HM, Scinto JM, Radford M. Warfarin use among patients with atrial fibrillation. Stroke. 1997 Dec;28(12):2382-9. doi: 10.1161/01.str.28.12.2382. PMID 9412618
- [Background] Go AS, Hylek EM, Borowsky LH, Phillips KA, Selby JV, Singer DE. Warfarin use among ambulatory patients with nonvalvular atrial fibrillation: the anticoagulation and risk factors in atrial fibrillation (ATRIA) study. Ann Intern Med. 1999 Dec 21;131(12):927-34. doi: 10.7326/0003-4819-131-12-199912210-00004. PMID 10610643
- [Background] Birman-Deych E, Radford MJ, Nilasena DS, Gage BF. Use and effectiveness of warfarin in Medicare beneficiaries with atrial fibrillation. Stroke. 2006 Apr;37(4):1070-4. doi: 10.1161/01.STR.0000208294.46968.a4. Epub 2006 Mar 9. PMID 16528001
- [Background] Mant J, Hobbs FD, Fletcher K, Roalfe A, Fitzmaurice D, Lip GY, Murray E; BAFTA investigators; Midland Research Practices Network (MidReC). Warfarin versus aspirin for stroke prevention in an elderly community population with atrial fibrillation (the Birmingham Atrial Fibrillation Treatment of the Aged Study, BAFTA): a randomised controlled trial. Lancet. 2007 Aug 11;370(9586):493-503. doi: 10.1016/S0140-6736(07)61233-1. PMID 17693178
- [Background] Broderick JP, Bonomo JB, Kissela BM, Khoury JC, Moomaw CJ, Alwell K, Woo D, Flaherty ML, Khatri P, Adeoye O, Ferioli S, Kleindorfer DO. Withdrawal of antithrombotic agents and its impact on ischemic stroke occurrence. Stroke. 2011 Sep;42(9):2509-14. doi: 10.1161/STROKEAHA.110.611905. Epub 2011 Jun 30. PMID 21719769
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Kalra L, Yu G, Perez I, Lakhani A, Donaldson N. Prospective cohort study to determine if trial efficacy of anticoagulation for stroke prevention in atrial fibrillation translates into clinical effectiveness. BMJ. 2000 May 6;320(7244):1236-9. doi: 10.1136/bmj.320.7244.1236. PMID 10797031
- [Background] Ono A, Fujita T. Low-intensity anticoagulation for stroke prevention in elderly patients with atrial fibrillation: efficacy and safety in actual clinical practice. J Clin Neurosci. 2005 Nov;12(8):891-4. doi: 10.1016/j.jocn.2004.10.011. Epub 2005 Nov 3. PMID 16271478
- [Background] Ruiz Ortiz M, Romo Penas E, Franco Zapata MF, Mesa Rubio D, Anguita Sanchez M, Lopez Granados A, Arizon del Prado JM, Valles Belsue F. Oral anticoagulation in patients aged 75 years or older with chronic non-valvar atrial fibrillation: effectiveness and safety in daily clinical practice. Heart. 2005 Sep;91(9):1225-6. doi: 10.1136/hrt.2004.050831. No abstract available. PMID 16103572
- [Background] Katz ES, Tsiamtsiouris T, Applebaum RM, Schwartzbard A, Tunick PA, Kronzon I. Surgical left atrial appendage ligation is frequently incomplete: a transesophageal echocardiograhic study. J Am Coll Cardiol. 2000 Aug;36(2):468-71. doi: 10.1016/s0735-1097(00)00765-8. PMID 10933359
- [Background] Holmes DR, Reddy VY, Turi ZG, Doshi SK, Sievert H, Buchbinder M, Mullin CM, Sick P; PROTECT AF Investigators. Percutaneous closure of the left atrial appendage versus warfarin therapy for prevention of stroke in patients with atrial fibrillation: a randomised non-inferiority trial. Lancet. 2009 Aug 15;374(9689):534-42. doi: 10.1016/S0140-6736(09)61343-X. PMID 19683639
- [Background] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Background] Holmes DR Jr, Doshi SK, Kar S, Price MJ, Sanchez JM, Sievert H, Valderrabano M, Reddy VY. Left Atrial Appendage Closure as an Alternative to Warfarin for Stroke Prevention in Atrial Fibrillation: A Patient-Level Meta-Analysis. J Am Coll Cardiol. 2015 Jun 23;65(24):2614-2623. doi: 10.1016/j.jacc.2015.04.025. PMID 26088300
- [Background] Reddy VY, Holmes D, Doshi SK, Neuzil P, Kar S. Safety of percutaneous left atrial appendage closure: results from the Watchman Left Atrial Appendage System for Embolic Protection in Patients with AF (PROTECT AF) clinical trial and the Continued Access Registry. Circulation. 2011 Feb 1;123(4):417-24. doi: 10.1161/CIRCULATIONAHA.110.976449. Epub 2011 Jan 17. PMID 21242484
- [Background] Price MJ, Reddy VY, Valderrabano M, Halperin JL, Gibson DN, Gordon N, Huber KC, Holmes DR Jr. Bleeding Outcomes After Left Atrial Appendage Closure Compared With Long-Term Warfarin: A Pooled, Patient-Level Analysis of the WATCHMAN Randomized Trial Experience. JACC Cardiovasc Interv. 2015 Dec 28;8(15):1925-1932. doi: 10.1016/j.jcin.2015.08.035. Epub 2015 Nov 25. PMID 26627989
- [Background] Boersma LV, Schmidt B, Betts TR, Sievert H, Tamburino C, Teiger E, Pokushalov E, Kische S, Schmitz T, Stein KM, Bergmann MW; EWOLUTION investigators. Implant success and safety of left atrial appendage closure with the WATCHMAN device: peri-procedural outcomes from the EWOLUTION registry. Eur Heart J. 2016 Aug;37(31):2465-74. doi: 10.1093/eurheartj/ehv730. Epub 2016 Jan 27. PMID 26822918
- [Background] Reddy VY, Mobius-Winkler S, Miller MA, Neuzil P, Schuler G, Wiebe J, Sick P, Sievert H. Left atrial appendage closure with the Watchman device in patients with a contraindication for oral anticoagulation: the ASAP study (ASA Plavix Feasibility Study With Watchman Left Atrial Appendage Closure Technology). J Am Coll Cardiol. 2013 Jun 25;61(25):2551-6. doi: 10.1016/j.jacc.2013.03.035. Epub 2013 Apr 10. PMID 23583249
- [Background] Main ML, Fan D, Reddy VY, Holmes DR, Gordon NT, Coggins TR, House JA, Liao L, Rabineau D, Latus GG, Huber KC, Sievert H, Wright RF, Doshi SK, Douglas PS. Assessment of Device-Related Thrombus and Associated Clinical Outcomes With the WATCHMAN Left Atrial Appendage Closure Device for Embolic Protection in Patients With Atrial Fibrillation (from the PROTECT-AF Trial). Am J Cardiol. 2016 Apr 1;117(7):1127-34. doi: 10.1016/j.amjcard.2016.01.039. Epub 2016 Feb 1. PMID 26993976
- [Background] Meincke F, Schmidt-Salzmann M, Kreidel F, Kuck KH, Bergmann MW. New technical and anticoagulation aspects for left atrial appendage closure using the WATCHMAN(R) device in patients not taking warfarin. EuroIntervention. 2013 Aug 22;9(4):463-8. doi: 10.4244/EIJV9I4A75. PMID 23965351
- [Background] Reddy VY, Doshi SK, Sievert H, Buchbinder M, Neuzil P, Huber K, Halperin JL, Holmes D; PROTECT AF Investigators. Percutaneous left atrial appendage closure for stroke prophylaxis in patients with atrial fibrillation: 2.3-Year Follow-up of the PROTECT AF (Watchman Left Atrial Appendage System for Embolic Protection in Patients with Atrial Fibrillation) Trial. Circulation. 2013 Feb 12;127(6):720-9. doi: 10.1161/CIRCULATIONAHA.112.114389. Epub 2013 Jan 16. PMID 23325525
- [Background] Fountain RB, Holmes DR, Chandrasekaran K, Packer D, Asirvatham S, Van Tassel R, Turi Z. The PROTECT AF (WATCHMAN Left Atrial Appendage System for Embolic PROTECTion in Patients with Atrial Fibrillation) trial. Am Heart J. 2006 May;151(5):956-61. doi: 10.1016/j.ahj.2006.02.005. No abstract available. PMID 16644311
- [Background] Gangireddy SR, Halperin JL, Fuster V, Reddy VY. Percutaneous left atrial appendage closure for stroke prevention in patients with atrial fibrillation: an assessment of net clinical benefit. Eur Heart J. 2012 Nov;33(21):2700-8. doi: 10.1093/eurheartj/ehs292. Epub 2012 Sep 24. PMID 23008509
- [Background] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Background] Lip GY, Frison L, Halperin JL, Lane DA. Identifying patients at high risk for stroke despite anticoagulation: a comparison of contemporary stroke risk stratification schemes in an anticoagulated atrial fibrillation cohort. Stroke. 2010 Dec;41(12):2731-8. doi: 10.1161/STROKEAHA.110.590257. Epub 2010 Oct 21. PMID 20966417
- [Background] Friberg L, Rosenqvist M, Lip GY. Evaluation of risk stratification schemes for ischaemic stroke and bleeding in 182 678 patients with atrial fibrillation: the Swedish Atrial Fibrillation cohort study. Eur Heart J. 2012 Jun;33(12):1500-10. doi: 10.1093/eurheartj/ehr488. Epub 2012 Jan 13. PMID 22246443
- [Background] Zhao Y, Herring AH, Zhou H, Ali MW, Koch GG. A multiple imputation method for sensitivity analyses of time-to-event data with possibly informative censoring. J Biopharm Stat. 2014;24(2):229-53. doi: 10.1080/10543406.2013.860769. PMID 24605967
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Applegate RJ, Yaqub M, Hermiller JB, Sood P, Yu S, Doostzadeh J, Williams JE, Farhat N, Caputo R, Lansky AJ, Cutlip DE, Sudhir K, Stone GW. Long-term (three-year) safety and efficacy of everolimus-eluting stents compared to paclitaxel-eluting stents (from the SPIRIT III Trial). Am J Cardiol. 2011 Mar 15;107(6):833-40. doi: 10.1016/j.amjcard.2010.10.069. Epub 2011 Jan 19. PMID 21247538
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Tzikas A, Holmes DR Jr, Gafoor S, Ruiz CE, Blomstrom-Lundqvist C, Diener HC, Cappato R, Kar S, Lee RJ, Byrne RA, Ibrahim R, Lakkireddy D, Soliman OI, Nabauer M, Schneider S, Brachman J, Saver JL, Tiemann K, Sievert H, Camm AJ, Lewalter T. Percutaneous left atrial appendage occlusion: the Munich consensus document on definitions, endpoints and data collection requirements for clinical studies. EuroIntervention. 2016 May 17;12(1):103-11. doi: 10.4244/EIJV12I1A18. PMID 27173870